CLINICAL TRIAL: NCT01209819
Title: Bone Mineral Density in Adults With Hyperphenylalaninemia
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Heather Saavedra, Clinical Instructor - Pediatrics, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-10-0262
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Phenylketonurias
Keywords: Bone Mineral Density; Adults
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hyperphenylalaninemia (HPA) is a rare metabolic disorder caused by a deficiency of the enzyme phenylalanine hydroxylase (PAH). Elevated plasma levels of phenylalanine (phe) cause mental retardation, microcephaly, delayed speech, seizures, eczema, and behavior problems. Adequate control of the plasma levels of phe by a phe-restricted diet can prevent the developmental and behavioral problems.

The foundation of this diet is a phe-free medical product/formula made from free amino acids. Based on longitudinal studies, it has been reported that the most benefit is attained by individuals who maintain a phe-restricted diet throughout life. Despite the obvious benefits of the diet, it has been suggested that the dietary restrictions may be associated with poor bone health in these patients. However, data supporting this has been reported in studies with small sample sizes and/or inadequate sample populations that include children. There is a paucity of data on bone health in adults with HPA.

The investigators propose an observational study to describe the bone health status among adults with a diagnosis of HPA and to compare them to established normative age and gender-specific values among healthy individuals. The investigators hypothesize that adults with HPA will have lower bone density as measured by a dual x-ray absorptiometry (DXA) scan compared to the established normative values.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HPA at birth
* Aged 18 or older

Exclusion Criteria:

* Peri-menopausal women
* Menopausal women
* Patients taking bisphosphonates
* Pregnant women
* Women who have been pregnant within one year of study enrollment
* Women who have breastfed within one year of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with PKU or benign HPA followed at The University of Texas Health Science Center at Houston will be invited to participate in the study. In addition, adults with PKU or benign HPA in the State of Texas will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather W Saavedra, MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States